CLINICAL TRIAL: NCT04345614
Title: Part 1: A Randomized Controlled Open-Label Study of CM4620 Injectable Emulsion (CM4620-IE) in Patients With Severe COVID-19 Pneumonia Part 2: A Randomized Double Blind, Placebo-Controlled Study of Auxora for the Treatment of Severe COVID-19 Pneumonia (CARDEA)
Brief Title: A Study of Auxora in Patients With Severe COVID-19 Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CalciMedica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM4620-204
Record Dates: First submitted 2020-04-07; First posted 2020-04-14 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Pneumonia
Keywords: COVID-19; Coronavirus; Pneumonia; Calcium release-activated calcium channel (CRAC) inhibitors; CM4620; Auxora
MeSH Terms: conditions — Pneumonia; COVID-19; Coronavirus Infections | interventions — zegocractin; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matching placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Auxora (Part 1) (Experimental): Patients were randomized 1:1 to receive either Auxora or standard of care
  Interventions: Drug: Auxora (Part 1)
- Standard of Care (Part 1) (Other): Patients were randomized 1:1 to receive either Auxora or standard of care
  Interventions: Drug: Standard of Care (Part 1)
- Auxora (Part 2) (Experimental): Patients were randomized 1:1 to receive Auxora or Placebo
  Interventions: Drug: Auxora (Part 2)
- Placebo (Part 2) (Placebo Comparator): Patients were randomized 1:1 to receive Auxora or Placebo
  Interventions: Drug: Placebo (Part 2)

INTERVENTIONS:
Drug: Auxora (Part 1) — Auxora will be given at 2.0 mg/kg (1.25 mL/kg) on Day 1 and then 1.6 mg/kg (1.0 mL/kg) on Days 2 and 3. All doses of Auxora will be administered intravenously (IV) over 4 hours.
  Other Names: CM4620-Injectable Emulsion (IE)
  Arms: Auxora (Part 1)
Drug: Standard of Care (Part 1) — Patients received standard of care
  Other Names: Placebo-Injectable Emulsion
  Arms: Standard of Care (Part 1)
Drug: Auxora (Part 2) — Auxora will be given at 2.0 mg/kg (1.25 mL/kg) on Day 1 and then 1.6 mg/kg (1.0 mL/kg) on Days 2 and 3. All doses of Auxora will be administered intravenously (IV) over 4 hours.
  Other Names: CM4620-Injectable Emulsion (IE)
  Arms: Auxora (Part 2)
Drug: Placebo (Part 2) — Placebo will be given at 2.0 mg/kg (1.25 mL/kg) on Day 1 and then 1.6 mg/kg (1.0 mL/kg) on Days 2 and 3. All doses of Placebo will be administered intravenously (IV) over 4 hours.
  Other Names: Placebo-Injectable Emulsion
  Arms: Placebo (Part 2)

SUMMARY:
Part 1 of this trial enrolled 30 patients to receive Auxora (formerly CM4620) in a 2:1 randomized, open label trial of patients with severe and critical COVID-19 pneumonia. Part 2 of this study randomized 284 patients and was a randomized, double blind, placebo-controlled (RCT) study that evaluated the efficacy, safety, and the pharmacokinetic profile of Auxora in patients with severe COVID-19 pneumonia. The number of patients with an imputed PaO2/FiO2 >200 randomized into the study was capped at 26. Another 258 patients with a PaO2/FiO2 ≤200 were enrolled. Patients with an estimated PaO2/FiO2 of 75-200 were stratified to ensure balanced randomization between the Auxora and placebo arms. Subgroup analyses were performed to explore how time to recovery is influenced by baseline variables and to evaluate the treatment effect at different levels of each of these variables. The dose of Auxora was 2.0 mg/kg (1.25 mL/kg) administered at 0 hour, and then 1.6 mg/kg (1 mL/kg) at 24 hours and 1.6 mg/kg (1 mL/kg) at 48 hours from the SFISD. The dose of placebo was 1.25 mL/kg administered at 0 hour and then 1 mL/kg at 24 hours and 1 mL/kg at 48 hours from the SFISD. Remdesivir, corticosteroids and convalescent plasma were allowed. The infusion of Auxora / Placebo started within 12 hours from the time the patient or LAR provided informed consent. Efficacy analyses will be presented by treatment group (Auxora vs Placebo) based on the Efficacy Analysis Set of the imputed PaO2/FiO2 ≤200 subgroup, except where it is specified otherwise. The statistical analysis approach was designed to assess the significance of the primary and first secondary endpoint using the Benjamini and Hochberg method to control the overall trial level alpha level.

ELIGIBILITY:
Part 1:

Inclusion Criteria

1. 1. The diagnosis of COVID-19 established standard RT-PCR assay;
2. At least 1 of the following symptoms:

   Fever, cough, sore throat, malaise, headache, muscle pain, dyspnea at rest or with exertion, confusion, or respiratory distress;
3. At least 1 of the following clinical signs:

   Respiratory rate ≥30, heart rate ≥125, SpO2 <93% on room air or requires >2L oxygen by nasal cannula to maintain SpO2 ≥93%, or PaO2/FiO2 <300, estimated from pulse oximetry or determined by arterial blood gas;
4. The presence of a respiratory infiltrate or abnormality consistent with pneumonia that is documented by either a CXR or CT scan of the lungs;
5. The patient is ≥18 years of age;
6. A female patient of childbearing potential must not attempt to become pregnant for 39 months, and if sexually active with a male partner, is willing to practice acceptable methods of birth control for 39 months after the last dose of CM4620-IE;
7. A male patient who is sexually active with a female partner of childbearing potential is willing to practice acceptable methods of birth control for 39 months after the last dose of CM4620-IE. A male patient must not donate sperm for 39 months;
8. The patient is willing and able to, or has a legal authorized representative (LAR) who is willing and able to, provide informed consent to participate, and to cooperate with all aspects of the protocol.

Exclusion Criteria:

1. Expected survival or time to withdrawal of life-sustaining treatments expected to be <7 days.
2. Do Not Intubate order;
3. Home mechanical ventilation (noninvasive ventilation or via tracheotomy) except for continuous positive airway pressure or bi-level positive airway pressure (CPAP/BIPAP) used solely for sleep-disordered breathing;
4. PaO2/FiO2 ≤75 at the time of Screening. The PaO2/FiO2 may be estimated from pulse oximetry (Appendix 1) or determined by arterial blood gas;
5. Noninvasive positive pressure ventilation;
6. Invasive mechanical ventilation via endotracheal intubation or tracheostomy;
7. ECMO;
8. Shock defined by the use of vasopressors;
9. Multiple organ dysfunction or failure;
10. Positive Influenza A or B testing if tested as local standard of care;
11. The patient has a history any of the following: Organ or hematologic transplant;HIV; Active hepatitis B, or hepatitis C infection;
12. Current treatment with:Chemotherapy; Immunosuppressive medications or immunotherapy at the time of consent; Hemodialysis or Peritoneal Dialysis
13. Have a history of venous thromboembolism (VTE) (deep vein thrombosis [DVT] or pulmonary embolism [PE]) within 12 weeks prior to screening or have a history of recurrent (> 1) VTE;
14. The patient is known to be pregnant or is nursing;
15. Currently participating in another study of an investigational drug or therapeutic medical device at the time of consent;
16. Allergy to eggs or any of the excipients in study drug.

Part 2:

Inclusion Criteria:

1. Has laboratory-confirmed SARS-CoV-2 infection as determined by polymerase chain reaction (PCR) or other commercial or public health assay in any specimen, as documented by either of the following:

   * PCR positive in sample collected < 72 hours prior to randomization;
   * PCR positive in sample collected ≥ 72 hours prior to randomization, with inability to obtain a repeat sample (e.g. due to lack of testing supplies, or limited testing capacity, or results taking >24 hours, etc.) or progressive disease suggestive of ongoing SARS-CoV-2 infection;
2. At least 1 of the following symptoms: Fever, cough, sore throat, malaise, headache, muscle pain, dyspnea at rest or with exertion, confusion, or respiratory distress;
3. At least 1 of the following signs at Screening or noted in the 24 hours before Screening:

   * PaO2/FiO2 ≤200 when receiving supplemental oxygen. The PaO2/FiO2 may be estimated from pulse oximetry (Appendix 1) or determined by arterial blood gas;
   * If SpO2 ≥97%, must be receiving 10L or more of supplemental oxygen;
4. The presence of a respiratory infiltrate or abnormality consistent with pneumonia that is documented by either a chest X-ray or computerized tomography scan of the lungs;
5. The patient is ≥ 18 years of age;
6. A female patient of childbearing potential must not attempt to become pregnant for 39 months, and if sexually active with a male partner, is willing to practice acceptable methods of birth control for 39 months after the last dose of CM4620-IE;
7. A male patient who is sexually active with a female partner of childbearing potential is willing to practice acceptable methods of birth control for 39 months after the last dose of CM4620-IE. A male patient must not donate sperm for 39 months;
8. The patient is willing and able to, or has a legal authorized representative (LAR) who is willing and able to, provide informed consent to participate, and to cooperate with all aspects of the protocol.

Exclusion Criteria:

1. Expected survival or time to withdrawal of life-sustaining treatments expected to be <7 days.
2. Do Not Intubate order;
3. Home mechanical ventilation (noninvasive ventilation or via tracheotomy) except for continuous positive airway pressure or bi-level positive airway pressure (CPAP/BIPAP) used solely for sleep-disordered breathing;
4. PaO2/FiO2 ≤75 at the time of Screening. The PaO2/FiO2 may be estimated from pulse oximetry (Appendix 1) or determined by arterial blood gas;
5. Noninvasive positive pressure ventilation;
6. Invasive mechanical ventilation via endotracheal intubation or tracheostomy;
7. Extracorporeal membrane oxygenation (ECMO);
8. Shock defined by the use of vasopressors;
9. Multiple organ dysfunction or failure;
10. Positive Influenza A or B testing if tested as local standard of care;
11. The patient has a history of any of the following: Organ or hematologic transplant; HIV; Active hepatitis B, or hepatitis C infection;
12. Current treatment with:Chemotherapy;Immunosuppressive medications or immunotherapy at the time of consent; c. Hemodialysis or Peritoneal Dialysis;
13. Have a history of venous thromboembolism (VTE) (deep vein thrombosis [DVT] or pulmonary embolism [PE]) within 12 weeks prior to screening or have a history of recurrent (> 1) VTE;
14. The patient is known to be pregnant or is nursing;
15. Currently participating in another study of an investigational drug or therapeutic medical device at the time of consent;
16. Allergy to eggs or any of the excipients in study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudarshan Hebbar, MD, Study Director — CalciMedica, Inc.
Locations (17):
- United States (17):
  - Long Beach Memorial, Long Beach, California
  - University of Southern California / LA County, Los Angeles, California
  - Sharp Memorial San Diego, San Diego, California
  - National Jewish Health / St. Joseph's Hospital, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - Baton Rouge General, Baton Rouge, Louisiana
  - Maine Medical Center, Portland, Maine
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Sinai Grace, Detroit, Michigan
  - Methodist Hospital, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Texas Tech University Medical Center, El Paso, Texas
  - John Peter Smith Hospital, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Aurora Baycare, Green Bay, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bruen C, Al-Saadi M, Michelson EA, Tanios M, Mendoza-Ayala R, Miller J, Zhang J, Stauderman K, Hebbar S, Hou PC. Auxora vs. placebo for the treatment of patients with severe COVID-19 pneumonia: a randomized-controlled clinical trial. Crit Care. 2022 Apr 8;26(1):101. doi: 10.1186/s13054-022-03964-8. PMID 35395943
- [Derived] Miller J, Bruen C, Schnaus M, Zhang J, Ali S, Lind A, Stoecker Z, Stauderman K, Hebbar S. Auxora versus standard of care for the treatment of severe or critical COVID-19 pneumonia: results from a randomized controlled trial. Crit Care. 2020 Aug 14;24(1):502. doi: 10.1186/s13054-020-03220-x. PMID 32795330
- See also: Related Info — http://link.springer.com/epdf/10.1186/s13054-022-03964-8?sharing_token=3Y8kSc8AgIpRHpdksMq6Im_BpE1tBhCbnbw3BuzI2RNgljyjp_MC0UeLOpYbVoy4Catf2o1CPvZ9wGTDZgUwpYZuWDT8bfuJG9TbOiKMNKveLI72hbHo2LeXuzTz9fRlS7nYiCG03iBRpWSw5DkjlyQVC7Vq2QJGkYrC6D_b6es=

RESULTS

PARTICIPANT FLOW:
Groups:
- Auxora (Part 1): Patients were randomized 2:1 to receive CM4620-IE or continue with the local standard of care.
  The dose of CM4620-IE was 2.0 mg/kg of CM4620-IE administered at 0 hour, and 1.6 mg/kg at 24 hours and 1.6 mg/kg at 48 hours
- Standard of Care (Part 1): Patients were randomized 2:1 to receive CM4620-IE or continue with the local standard of care.
- Auxora (Part 2): Patients will be randomized 1:1 to receive either Auxora or placebo
  Auxora: Auxora will be given at 2.0 mg/kg (1.25 mL/kg) on Day 1 and then 1.6 mg/kg (1.0 mL/kg) on Days 2 and 3. All doses of Auxora will be administered intravenously (IV) over 4 hours.
- Placebo (Part 2): Patients will be randomized 1:1 to receive either Auxora or placebo
  Placebo: Placebo will be given at 1.25 mL/kg on Day 1 and then 1.0 mL/kg on Days 2 and 3. All doses of placebo will be administered intravenously over 4 hours.
Period: Overall Study
Arm/Group | Auxora (Part 1) | Standard of Care (Part 1) | Auxora (Part 2) | Placebo (Part 2)
Started | 20 | 10 | 143 | 141
Part 1: Low -Flow Oxygen Therapy Part 2: PaO2/FiO2 </= 200 | 17 (Of the 20 patients randomized to the Auxora arm, 17 of the patients were on low flow oxygen therapy and part of the pre-identified efficacy set.) | 9 (Of the 10 patients randomized to the standard of care arm, 9 were on low flow oxygen therapy and part of the pre-identified efficacy set) | 130 (Of the 143 patients, 130 patients with imputed PaO2/FiO2 </= 200 were randomized to this group and part of the pre-identified efficacy set.) | 131 (Of the 143 patients, 131 patients with imputed PaO2/FiO2 </= 200 were randomized to this group and part of the pre-identified efficacy set.)
Completed | 20 | 10 | 143 | 141
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Auxora (Part 2): Patients were randomized 1:1 to receive either Auxora or placebo
  Auxora: Auxora was given at 2.0 mg/kg (1.25 mL/kg) on Day 1 and then 1.6 mg/kg (1.0 mL/kg) on Days 2 and 3. All doses of Auxora will be administered intravenously (IV) over 4 hours.
- Placebo (Part 2): Patients were randomized 1:1 to receive either Auxora or placebo
  Placebo: Placebo was given at 1.25 mL/kg on Day 1 and then 1.0 mL/kg on Days 2 and 3. All doses of placebo will be administered intravenously over 4 hours.
- Total: Total of all reporting groups
Arm/Group | Auxora (Part 1) | Standard of Care (Part 1) | Auxora (Part 2) | Placebo (Part 2) | Total
Number analyzed (Participants) | 17 | 9 | 130 | 131 | 287
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: For Part 1 of the study, all 30 treated patients were included in the MITT population, and 26 patients in the low-flow (severe COVID-19 pneumonia) arm were included in the efficacy evaluable population.In Part 2, 261 patients (131 placebo and 130 Auxora patients) with a baseline imputed PaO2/FiO2 ≤200 group were included in the Efficacy Analysis Set 281 patients (140 placebo and 141 Auxora patients) were included in the Safety Analysis Set
  years | 59.3 (12.47) | 61.0 (13.32) | 59.4 (12.1) | 60.4 (12.3) | 59.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: For Part 1 of the study, all 30 treated patients were included in the MITT population, and 26 patients in the low-flow (severe COVID-19 pneumonia) arm were included in the efficacy evaluable population.In Part 2, 261 patients (131 placebo and 130 Auxora patients) with a baseline imputed PaO2/FiO2 ≤200 group were included in the Efficacy Analysis Set 281 patients (140 placebo and 141 Auxora patients) were included in the Safety Analysis Set
  Participants
    Female | 10 | 4 | 46 | 39 | 99
    Male | 7 | 5 | 84 | 92 | 188
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 45 | 58 | 106
  Not Hispanic or Latino | 14 | 6 | 82 | 72 | 174
  Unknown or Not Reported | 1 | 2 | 3 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants] — Category "More than one race" also includes patients who indicated "other"
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 1 | 9 | 5 | 15
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
    Black or African American | 7 | 3 | 19 | 12 | 41
    White | 8 | 5 | 85 | 98 | 196
    More than one race | 2 | 0 | 16 | 15 | 33
    Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 17 | 9 | 130 | 131 | 287
65+years of age [Count of Participants; unit: Participants] — Population: For Part 1 of the study, all 30 treated patients were included in the MITT population, and 26 patients in the low-flow (severe COVID-19 pneumonia) arm were included in the efficacy evaluable population.In Part 2, 261 patients (131 placebo and 130 Auxora patients) with a baseline imputed PaO2/FiO2 ≤200 group were included in the Efficacy Analysis Set 281 patients (140 placebo and 141 Auxora patients) were included in the Safety Analysis Set
  Participants | 4 | 4 | 45 | 47 | 100
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: For Part 1 of the study, all 30 treated patients were included in the MITT population, and 26 patients in the low-flow (severe COVID-19 pneumonia) arm were included in the efficacy evaluable population.In Part 2, 261 patients (131 placebo and 130 Auxora patients) with a baseline imputed PaO2/FiO2 ≤200 group were included in the Efficacy Analysis Set 281 patients (140 placebo and 141 Auxora patients) were included in the Safety Analysis Set
  kg/m^2 | 34.4 (13.5) | 33.1 (8.58) | 32.8 (8.8) | 32.0 (7.0) | 32.4 (8.0)
Time from symptom onset [Mean (Standard Deviation); unit: Days] — Population: For Part 1 of the study, all 30 treated patients were included in the MITT population, and 26 patients in the low-flow (severe COVID-19 pneumonia) arm were included in the efficacy evaluable population.In Part 2, 261 patients (131 placebo and 130 Auxora patients) with a baseline imputed PaO2/FiO2 ≤200 group were included in the Efficacy Analysis Set 281 patients (140 placebo and 141 Auxora patients) were included in the Safety Analysis Set
  Days | 11.1 (7.13) | 6.9 (2.59) | 12.2 (5.8) | 12.0 (5.9) | 12.1 (5.8)
High-flow nasal cannula use (HFNC) [Count of Participants; unit: Participants] — Population: For Part 1 of the study, all 30 treated patients were included in the MITT population, and 26 patients in the low-flow (severe COVID-19 pneumonia) arm were included in the efficacy evaluable population.In Part 2, 261 patients (131 placebo and 130 Auxora patients) with a baseline imputed PaO2/FiO2 ≤200 group were included in the Efficacy Analysis Set 281 patients (140 placebo and 141 Auxora patients) were included in the Safety Analysis Set
  Participants | 0 | 0 | 81 | 82 | 163
Baseline imputed PaO2/FiO2 value [Mean (Standard Deviation); unit: Ratio] — Population: For Part 1 of the study, all 30 treated patients were included in the MITT population, and 26 patients in the low-flow (severe COVID-19 pneumonia) arm were included in the efficacy evaluable population.In Part 2, 261 patients (131 placebo and 130 Auxora patients) with a baseline imputed PaO2/FiO2 ≤200 group were included in the Efficacy Analysis Set 281 patients (140 placebo and 141 Auxora patients) were included in the Safety Analysis Set
  Ratio | 177.5 (74.03) | 167.6 (77.60) | 109.7 (36.8) | 105.1 (32.8) | 107.4 (34.8)
Baseline imputed PaO2/FiO2=/<100 [Count of Participants; unit: Participants] — Population: For Part 1 of the study, all 30 treated patients were included in the MITT population, and 26 patients in the low-flow (severe COVID-19 pneumonia) arm were included in the efficacy evaluable population.In Part 2, 261 patients (131 placebo and 130 Auxora patients) with a baseline imputed PaO2/FiO2 ≤200 group were included in the Efficacy Analysis Set 281 patients (140 placebo and 141 Auxora patients) were included in the Safety Analysis Set
  Participants | 4 | 2 | 59 | 58 | 123
Baseline imputed PaO2/FiO2 101-200 [Count of Participants; unit: Participants] — Population: For Part 1 of the study, all 30 treated patients were included in the MITT population, and 26 patients in the low-flow (severe COVID-19 pneumonia) arm were included in the efficacy evaluable population.In Part 2, 261 patients (131 placebo and 130 Auxora patients) with a baseline imputed PaO2/FiO2 ≤200 group were included in the Efficacy Analysis Set 281 patients (140 placebo and 141 Auxora patients) were included in the Safety Analysis Set
  Participants | 6 | 4 | 71 | 73 | 154
C-reactive protein (CRP) [Mean (Standard Deviation); unit: mg/L] — Population: For Part 1 of the study, all 30 treated patients were included in the MITT population, and 26 patients in the low-flow (severe COVID-19 pneumonia) arm were included in the efficacy evaluable population.In Part 2, 261 patients (131 placebo and 130 Auxora patients) with a baseline imputed PaO2/FiO2 ≤200 group were included in the Efficacy Analysis Set 281 patients (140 placebo and 141 Auxora patients) were included in the Safety Analysis Set
  mg/L | 99.9 (68.34) | 124.3 (59.28) | 93.1 (71.2) | 92.5 (67.6) | 92.8 (69.2)
Ferritin [Mean (Standard Deviation); unit: ng/mL] — Population: For Part 1 of the study, all 30 treated patients were included in the MITT population, and 26 patients in the low-flow (severe COVID-19 pneumonia) arm were included in the efficacy evaluable population.In Part 2, 261 patients (131 placebo and 130 Auxora patients) with a baseline imputed PaO2/FiO2 ≤200 group were included in the Efficacy Analysis Set 281 patients (140 placebo and 141 Auxora patients) were included in the Safety Analysis Set
  ng/mL | 709.1 (553.09) | 771.6 (741.57) | 1027 (907) | 1050 (869) | 1039 (886)
Hypertension [Count of Participants; unit: Participants] — Population: For Part 1 of the study, all 30 treated patients were included in the MITT population, and 26 patients in the low-flow (severe COVID-19 pneumonia) arm were included in the efficacy evaluable population.In Part 2, 261 patients (131 placebo and 130 Auxora patients) with a baseline imputed PaO2/FiO2 ≤200 group were included in the Efficacy Analysis Set 281 patients (140 placebo and 141 Auxora patients) were included in the Safety Analysis Set
  Participants | 8 | 4 | 84 | 80 | 176
Diabetes [Count of Participants; unit: Participants] — Population: For Part 1 of the study, all 30 treated patients were included in the MITT population, and 26 patients in the low-flow (severe COVID-19 pneumonia) arm were included in the efficacy evaluable population.In Part 2, 261 patients (131 placebo and 130 Auxora patients) with a baseline imputed PaO2/FiO2 ≤200 group were included in the Efficacy Analysis Set 281 patients (140 placebo and 141 Auxora patients) were included in the Safety Analysis Set
  Participants | 8 | 2 | 52 | 57 | 119
Hyperlipidemia [Count of Participants; unit: Participants] — Population: For Part 1 of the study, all 30 treated patients were included in the MITT population, and 26 patients in the low-flow (severe COVID-19 pneumonia) arm were included in the efficacy evaluable population.In Part 2, 261 patients (131 placebo and 130 Auxora patients) with a baseline imputed PaO2/FiO2 ≤200 group were included in the Efficacy Analysis Set 281 patients (140 placebo and 141 Auxora patients) were included in the Safety Analysis Set
  Participants | 2 | 0 | 50 | 51 | 103
Former smoker [Count of Participants; unit: Participants] — Population: For Part 1 of the study, all 30 treated patients were included in the MITT population, and 26 patients in the low-flow (severe COVID-19 pneumonia) arm were included in the efficacy evaluable population.In Part 2, 261 patients (131 placebo and 130 Auxora patients) with a baseline imputed PaO2/FiO2 ≤200 group were included in the Efficacy Analysis Set 281 patients (140 placebo and 141 Auxora patients) were included in the Safety Analysis Set
  Participants | 5 | 2 | 39 | 34 | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Days From the Start of the First Infusion of Study Drug (SFISD) to Recovery
Description: Defined as the number of days hospitalized but not requiring supplemental oxygen or ongoing medical care, or; discharged and requiring supplemental oxygen, or; discharged, not requiring supplemental oxygen.
Time Frame: From start of first infusion of study drug to day 60
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Auxora (Part 2): Patients were randomized 1:1 to receive either Auxora or placebo
  Auxora: Auxora was given at 2.0 mg/kg (1.25 mL/kg) on Day 1 and then 1.6 mg/kg (1.0 mL/kg) on Days 2 and 3. All doses of Auxora were administered intravenously (IV) over 4 hours.
Arm/Group | Auxora (Part 1) | Standard of Care (Part 1) | Auxora (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 17 | 9 | 130 | 131
Days | 5 [3.0 to 10] | 12 [2.0 to 12] | 7.0 [6.0 to 9.0] | 10.0 [7.0 to 14.0]

2. Secondary Outcome: Number of Participants Who Have Died at Day 30 (Mortality)
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Auxora (Part 1) | Standard of Care (Part 1) | Auxora (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 17 | 9 | 130 | 131
Participants | 2 | 2 | 10 | 23

3. Secondary Outcome: Number of Participants Who Have Died at Day 60 (Mortality)
Time Frame: Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Auxora (Part 1) | Standard of Care (Part 1) | Auxora (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 17 | 9 | 130 | 131
Participants | 2 | 2 | 18 | 27

4. Secondary Outcome: Number of Participants Requiring Invasive Mechanical Ventilation or Dying (Part 1)
Time Frame: From start of first infusion of study drug and up to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Auxora (Part 1) | Standard of Care (Part 1)
Number analyzed (Participants) | 17 | 9
Participants | 4 | 5

5. Secondary Outcome: Proportion of Patients Requiring Invasive Mechanical Ventilation or Dying (Part 2)
Time Frame: from start of first infusion of study drug and up to day day 60
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Auxora (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 130 | 131
Proportion of Participants | .23 [0.17 to 0.31] | .31 [0.24 to 0.39]

6. Secondary Outcome: Proportion of Patients Requiring Invasive Mechanical Ventilation (Part 2)
Time Frame: from start of first infusion of study drug and up to day Day 60
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Auxora (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 130 | 131
Proportion of participants | 0.19 [0.13 to 0.28] | 0.28 [0.21 to 0.37]

7. Secondary Outcome: Improvement in 8-point Ordinal Scale (Part 1)
Description: The ordinal scale is an assessment of the clinical status in a given day. The scale is as follows: 1. Death 2. Hospitalized, requiring invasive mechanical ventilation or ECMO 3. Hospitalized, requiring non-invasive ventilation or high flow supplemental oxygen 4. Hospitalized, requiring low flow supplemental oxygen 5. Hospitalized, not requiring supplemental oxygen, but requiring ongoing medical care 6. Hospitalized, not requiring supplemental oxygen or ongoing medical care 7. discharged, requiring supplemental oxygen 8. Discharged, not requiring supplemental oxygen
Time Frame: from start of first infusion of study drug and up to day 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Auxora (Part 1) | Standard of Care (Part 1)
Number analyzed (Participants) | 17 | 9
score on a scale | 6.3 (2.39) | 4.6 (2.92)

8. Secondary Outcome: Differences in Outcomes as Measured by an 8-point Ordinal Scale (Part 2)
Description: as for outcome 7
Time Frame: from start of first infusion of study drug hrough Day 60
Measure: Count of Participants; unit: Participants
Groups:
- Auxora Baseline; Auxora Day 12; Auxora Day 30; Auxora Day 60: Patients will be randomized 1:1 to receive either Auxora or placebo
  Auxora: Auxora will be given at 2.0 mg/kg (1.25 mL/kg) on Day 1 and then 1.6 mg/kg (1.0 mL/kg) on Days 2 and 3. All doses of Auxora will be administered intravenously (IV) over 4 hours.
- Placebo Baseline; Placebo Day 12; Placebo Day 30; Placebo Day 60: Patients will be randomized 1:1 to receive either Auxora or placebo
  Placebo: Placebo will be given at 1.25 mL/kg on Day 1 and then 1.0 mL/kg on Days 2 and 3. All doses of placebo will be administered intravenously over 4 hours.
Arm/Group | Auxora Baseline | Placebo Baseline | Auxora Day 12 | Placebo Day 12 | Auxora Day 30 | Placebo Day 30 | Auxora Day 60 | Placebo Day 60
Number analyzed (Participants) | 130 | 131 | 122 | 129 | 124 | 129 | 124 | 129
Participants
  1 | 0 | 0 | 5 | 8 | 10 | 23 | 18 | 27
  2 | 0 | 0 | 11 | 23 | 11 | 8 | 3 | 5
  3 | 81 | 82 | 17 | 16 | 5 | 3 | 0 | 0
  4 | 49 | 49 | 6 | 7 | 2 | 2 | 0 | 0
  5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  6 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 5
  7 | 0 | 0 | 38 | 39 | 24 | 33 | 32 | 33
  8 | 0 | 0 | 45 | 36 | 71 | 58 | 69 | 59

9. Secondary Outcome: Change in PaO2/FiO2 (Part 1)
Description: Measures of PaO2/FiO2 ratio
Time Frame: From start of first infusion of study drug through Day 28
Measure: Mean (Standard Deviation); unit: ratio of the arterial partial pressure o
Arm/Group | Auxora (Part 1) | Standard of Care (Part 1)
Number analyzed (Participants) | 17 | 9
ratio of the arterial partial pressure o | 66.94 (152.673) | 153.31 (153.258)

10. Secondary Outcome: Number of Days in the Hospital(Part 1)
Description: Time to discharge alive from hospital
Time Frame: From start of first infusion of study drug through Discharge up to 28 days
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Auxora (Part 1) | Standard of Care (Part 1)
Number analyzed (Participants) | 17 | 9
Days | 5 [3 to 10] | 12 [2 to NA] — Not enough events to determine upper CI value

11. Secondary Outcome: Number of Days in the Hospital (Part 2)
Time Frame: from admission into the hospital until discharge from the hospital up to 60 days
Population: Number of days in the hospital during the first 28 days of the study with a baseline imputed PaO2/FiO2 </= 200
Measure: Least Squares Mean (95% Confidence Interval); unit: Days
Groups:
- Auxora: Patients will be randomized 1:1 to receive either Auxora or placebo
  Auxora: Auxora will be given at 2.0 mg/kg (1.25 mL/kg) on Day 1 and then 1.6 mg/kg (1.0 mL/kg) on Days 2 and 3. All doses of Auxora will be administered intravenously (IV) over 4 hours.
- Placebo: Patients will be randomized 1:1 to receive either Auxora or placebo
  Placebo: Placebo will be given at 1.25 mL/kg on Day 1 and then 1.0 mL/kg on Days 2 and 3. All doses of placebo will be administered intravenously over 4 hours.
Arm/Group | Auxora | Placebo
Number analyzed (Participants) | 130 | 131
Days | 13.65 [11.92 to 15.38] | 15.29 [13.57 to 17.01]

12. Secondary Outcome: Number of Days in the Intensive Care Unit (ICU) (Part 2)
Time Frame: from admission into ICU until discharge from ICU up to 60 days
Population: Number of ICU days during the first 28 days of the study in patients with a baseline imputed PaO2/FiO2 </= 200
Measure: Least Squares Mean (Inter-Quartile Range); unit: Days
Arm/Group | Auxora | Placebo
Number analyzed (Participants) | 130 | 131
Days | 6.88 [4.92 to 8.85] | 8.36 [6.40 to 10.32]

13. Secondary Outcome: Days Alive and Free of Mechanical Ventilation (Part 1)
Time Frame: From randomization through Day 28
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Auxora (Part 1) | Standard of Care (Part 1)
Number analyzed (Participants) | 17 | 9
Days | 22.9 (10.3) | 12.9 (14.3)

14. Secondary Outcome: Number of Participants Considered Recovered (Part 1)
Description: Recovery is defined as a 6, 7, or 8 on the 8 point ordinal scale
Time Frame: From start of first infusion of study drug through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Auxora (Part 1) | Standard of Care (Part 1)
Number analyzed (Participants) | 17 | 9
Participants | 14 | 4

15. Secondary Outcome: CM4620-IE Plasma Concentration (Part 2)
Description: Concentration measured using a validated assay
Time Frame: From start of first infusion of study drug through 72 hours
Population: Patients with a viable PK sample at 72 hours
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Auxora | Placebo
Number analyzed (Participants) | 71 | 0
ng/mL | 165.2 (91.9) |

16. Secondary Outcome: Percentage of Patients With Treatment Emergent Adverse Events (TEAE) and Serious Adverse Events (SAE)
Time Frame: From start of first infusion of study drugand through day 60
Population: For Part 1 of the study, all 30 treated patients were included in the Safety Analysis Set. In Part 2, 281 patients (140 placebo and 141 Auxora patients) were included in the Safety Analysis Set
Measure: Number; unit: percentage of patients
Arm/Group | Auxora (Part 1) | Standard of Care (Part 1) | Auxora (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 20 | 10 | 141 | 140
percentage of patients
  Patients with at least 1 TEAE | 75.0 | 80.0 | 64.5 | 61.4
  Mild TEAE | 20.0 | 20.0 | 29.8 | 17.9
  Moderate TEAE | 25.0 | 10.0 | 10.6 | 8.6
  Severe TEAE | 25.0 | 10.0 | 24.1 | 35
  Patients with at least one treatment related TEAE | 15.0 | 0.0 | 25.5 | 12.9

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected from randomization through Day 60
Arm/Group | Auxora (Part 1) | Standard of Care (Part 1) | Auxora (Part 2) | Placebo (Part 2)
All-Cause Mortality (participants affected / at risk) | 2/20 | 2/10 | 18/141 | 27/140
Serious Adverse Events (participants affected / at risk) | 6/20 | 5/10 | 34/141 | 49/140
Other Adverse Events (participants affected / at risk) | 15/20 | 8/10 | 69/141 | 68/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Auxora (Part 1) (N=20) | Standard of Care (Part 1) (N=10) | Auxora (Part 2) (N=141) | Placebo (Part 2) (N=140)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 2 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 6 | 6
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Conduction Disorder (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary Artery Occlusion (Cardiac disorders) | 0 | 0 | 0 | 1
Pulseless Electrical Activity (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Bacterial Pneumonia (Infections and infestations) | 2 | 0 | 1 | 0
Klebsiella Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 6 | 7
Pneumonia Klebsiella (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia Staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1
Pseudomonal Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Septic shock (Infections and infestations) | 3 | 2 | 2 | 8
Staphylococcal Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0
Decreased Oxygen Saturation (Investigations) | 0 | 0 | 1 | 0
Increased Liver Function Test (Investigations) | 0 | 0 | 0 | 1
Brain Injury (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 1 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 2 | 4
ARDS (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 7 | 11
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 2
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 2
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 22 | 26
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 2 | 3
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Shock (Vascular disorders) | 1 | 0 | 2 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Auxora (Part 1) (N=20) | Standard of Care (Part 1) (N=10) | Auxora (Part 2) (N=141) | Placebo (Part 2) (N=140)
Blood triglycerides increased (Metabolism and nutrition disorders) | 1 | 2 | 16 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 0 | 11 | 11
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 8 | 12
Increased transaminases (Investigations) | 0 | 0 | 8 | 5
DVT (Vascular disorders) | 0 | 1 | 5 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 4 | 6
Anemia (Blood and lymphatic system disorders) | 2 | 1 | 2 | 8
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 3
Blood Alkaline Phosphatase Increased (Investigations) | 2 | 0 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 2 | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 1 | 2 | 1
Abdominal Pain (General disorders) | 0 | 1 | 4 | 2
Chills (General disorders) | 0 | 1 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 2 | 3
Decubitus Ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 1 | 2
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 2
Normocytic Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The number of patients who participated in the biomarker collection was not sufficient to provide / record meaningful results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/14/NCT04345614/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT04345614/SAP_001.pdf